CLINICAL TRIAL: NCT02583698
Title: Efficacy of Nonselective Beta Blockers vs Placebo in Patients With Acute-on-chronic Liver Failure With Small/ no Esophageal Varices
Brief Title: Efficacy of Nonselective Beta Blocker vs Placebo in Patients With Acute-on-chronic Liver Failure With Small/ no Esophageal Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-005
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2017-11

CONDITIONS: Acute on Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure | interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Tab Carvedilol 3.125 mg twice daily followed by 6.25 mg BD and finally 12.5 mg BD if SBP > 90 mmHg and HR >55/min
  Interventions: Drug: Carvedilol
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Carvedilol
  Arms: Carvedilol
Drug: Placebo
  Arms: placebo

SUMMARY:
Acute on chronic liver failure patients with HVPG (Hepatic Venous Pressure Gradient) ≥ 12 mmHg + No/small esophageal varices who present to the Department of Hepatology at Institute of Liver and Billiary Sciences, who meet the inclusion criteria and who provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Acute on Chronic Liver Failure as per APASL (Asian Pacific Association of Study of Liver Disease) criteria.
2. 18-75 years
3. HVPG ≥ 12 + No/Small Esophageal varices

Exclusion Criteria:

1. Bradycardia (HR < 60/ min)
2. Hypotension
3. Asthma
4. LVF
5. AKI (Acute Kidney Injury), (S.creat >1.5)
6. Refractory ascites
7. SBP (Spontaneous Bacterial Peritonitis)
8. Pregnancy or Lactation
9. Past history of EVL or EST
10. Significant cardio - pulmonary co-morbidity
11. PVT
12. Presence of grades 3-4 hepatic encephalopathy (HE)
13. Patients going for liver transplant in next 12 weeks
14. No consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Mortality in both groups | 28 days

SECONDARY OUTCOMES:
Number of patients with development or progression of esophageal varices in both groups. | 3 Months
Number of patients with reduction in hepatic venous pressure gradient (HVPG) in both groups. | 3 Months
Number of patients with regression in esophageal varices in both groups. | 3 Months
Number of patients with improvement in Liver severity scores in both groups. | 28 days
Number of patients with improvement in Liver severity scores in both groups. | 60 days
Number of patients with improvement in Liver severity scores in both groups. | 3 months
Number of patients with development of adverse events in both groups in both groups. | 28 days
Number of patients with development of adverse events in both groups in both groups. | 2 months
Number of patients with development of adverse events in both groups in both groups. | 3 Months
Number of patients who will develop esophageal variceal bleeding in both groups | 28 days
Number of patients who will develop esophageal variceal bleeding in both groups | 2 Months
Number of patients who will develop esophageal variceal bleeding in both groups | 3 Months
Development of complications in both groups | 28 days
  AKI,Pneumonia,SBP and other infections
Development of complications in both groups | 2 months
  AKI,Pneumonia,SBP and other infections
Development of complications in both groups | 3 months
  AKI,Pneumonia,SBP and other infections
Mortality in both groups | 2 months
Mortality in both groups | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Sumeet Kainth, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kumar M, Kainth S, Choudhury A, Maiwall R, Mitra LG, Saluja V, Agarwal PM, Shasthry SM, Jindal A, Bhardwaj A, Kumar G, Sarin SK. Treatment with carvedilol improves survival of patients with acute-on-chronic liver failure: a randomized controlled trial. Hepatol Int. 2019 Nov;13(6):800-813. doi: 10.1007/s12072-019-09986-9. Epub 2019 Sep 20. PMID 31541422